CLINICAL TRIAL: NCT05893771
Title: Evaluation of the Feasibility of Depomedrol Added to Bupivacaine in Ultrasound-guided Genicular Nerve Block in the Combination With Adductor Canal Block for Postoperative Analgesia and Rehabilitation After Reconstructive Knee Surgery.
Brief Title: Depomedrol for Genicular Nerve Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hazem Ezzat Elsersy, assistant professor of anesthesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4/2023ANET16
Record Dates: First submitted 2023-05-16; First posted 2023-06-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Methylprednisolone; Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will be allocated into three equal parallel groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, caregivers, investigators, and outcome assessors will be blinded by a pharmacist who will prepare medications in colorless coded sterile syringes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo control (Placebo Comparator): With ultrasound guidance, 20 ml plain normal saline will be injected to spread lateral to the femoral artery and deep to the sartorius muscle, or more distal, below the knee after arrival to the theatre.
  Interventions: Drug: normal saline
- Depomedrol group (Experimental): With ultrasound guidance, a mixture of 5 ml Bupivacaine 0.5%, 1 ml (20 mg) depomedrol, and 14 ml normal saline is injected to spread lateral to the femoral artery and deep to the sartorius muscle, or more distal, below the knee after arrival at the theatre.
  Interventions: Drug: Methylprednisolone Injection; Drug: Bupivacaine Hcl 0.5% Inj_#2; Drug: normal saline
- Bupivacaine group (Active Comparator): A mixture of 5 ml Bupivacaine 0.5%- and 14-ml normal saline is injected to spread lateral to the femoral artery and deep to the sartorius muscle, or more distal, below the knee, after arrival at the theatre.
  Interventions: Drug: Bupivacaine Hcl 0.5% Inj_#2; Drug: normal saline

INTERVENTIONS:
Drug: Methylprednisolone Injection — Ultrasound-guided genicular nerve block comparing Methylprednisolone combined with Bupivacaine to bupivacaine alone. All patients will undergo TKA and will receive spinal anesthesia.
  Other Names: Depomedrol
  Arms: Depomedrol group
Drug: Bupivacaine Hcl 0.5% Inj_#2 — Ultasound- guided genicular nerve block using 5 ml bupivacaine 0.5% in 15 ml saline
  Other Names: Marcaine 0.5%
  Arms: Bupivacaine group; Depomedrol group
Drug: normal saline — Ultrasound guided genicular nerve infiltration with 20 ml normal saline as a placebo control.
  Other Names: 0.9% saline

SUMMARY:
This study is designed to test the efficacy of adding Depomedrol a long-acting steroid to bupivacaine for relieving postoperative pain and reducing opioid requirements following total knee replacement surgery. For this purpose, Depomedrol will be added to bupivacaine for ultrasound-guided Genicular nerve block combined with spinal anesthesia.

DETAILED DESCRIPTION:
TKA remains a challenge for physicians as more than half of these patients experience extreme knee pain immediately after surgery. The management of pain in patients undergoing total knee arthroplasty (TKA) remains a challenge for the anesthesiologist even with regional anesthesia as no single regional technique is adequate to balance effective analgesia with minimal muscle weakness. Severe postoperative pain following TKA has been shown to negatively affect early mobilization, physical rehabilitation, time to discharge, and overall post-op recovery. Multimodal analgesia incorporating regional anesthesia techniques provides optimum analgesia and minimizes the use of opioids and their side effects. Proximal nerve blocks such as the lumbar plexus, femoral nerve, and proximal sciatic nerve blocks provide excellent analgesia but frequently cause motor weakness, which reduces the patient's mobility. A distal blockade of genicular branches has also been described using ultrasound in acute and chronic pain management with fewer side effects. The superior medial genicular nerve and lateral genicular nerve can be identified using ultrasound and blocked at the level of the medial intramuscular, and lateral femoral epicondyles deep to the vastus medialis and lateralis, respectively. The inferior medial genicular nerve can be also targeted medial to the tibial plateau adjacent to the genicular vessels. Methylprednisolone acetate (MPA)(Depomedrol) is a lipophilic glucocorticoid commonly used in chronic pain procedures. It has a good safety record and its analgesic action can last from days to weeks.(8) The literature supporting its role as an adjuvant to local anesthetic in peripheral nerve block are scanty. However, some studies showed that depo-methylprednisolone as an adjuvant to 0.5% lidocaine showed excellent results in neuropathic pain resulting from nerve injury. This study aims to evaluate the efficacy of adding depomedrol as an additive to bupivacaine in genicular nerve block for evaluating postoperative pain, opioid use, and ease of ambulation in patients undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for primary elective total knee arthroplasty.
* American Society of Anesthesiologists Physical Status I-III.
* BMI 18-35 kg/m2.

Exclusion Criteria:

* Bleeding disorders.
* Allergy to any of the drugs used in the study.
* Renal insufficiency.
* Liver failure
* Neurological abnormalities (uncooperative or psychologically unstable patients).
* Patient refusal.
* Contraindication to a peripheral nerve block.
* ASA IV or V.
* Skin lesions/infection at block site.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours.
  will be assessed postoperatively using 10 points numerical rating scale (NRS) where 0 no pain and 10 is the most intense pain. The median of pain scores through 48 hours will be compared.

SECONDARY OUTCOMES:
Opioid consumption | 24 hours, 48 hours.
  The amounts of Morphine in milligrams required by each patient will be recorded and compared.
Ambulation distance | Day one, day2 and day3
  The distance in meters that every patient can move without stopping pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all of the individual participant data collected during the trial after deidentification.
Supporting Information: Study Protocol
Time Frame: After 6 months from publication date and for 5 years